CLINICAL TRIAL: NCT06247956
Title: A Randomized, Open, Multicenter Phase II Clinical Study of SHR-8068 Combined With Adebrelimab and Platinum-containing Chemotherapy in the First-line Treatment of Advanced Gastric and Esophageal Cancer
Brief Title: Study of SHR-8068 Combined With Adebrelimab and Platinum-containing Chemotherapy in the Treatment of Advanced Gastric and Esophageal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SHR-8068-201-GC
Record Dates: First submitted 2024-01-30; First posted 2024-02-08 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Advanced Gastric Adenocarcinoma and Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-8068 combined with adebrelimab and platinum-containing chemotherapy (Experimental)
  Interventions: Drug: SHR-8068;Adebrelimab;Oxaliplatin;Capecitabine Tablets;Paclitaxel Injection;Cisplatin Injection
- Adebrelimab combined with platinum-containing chemotherapy (Active Comparator)
  Interventions: Drug: Adebrelimab;Oxaliplatin;Capecitabine Tablets;Paclitaxel Injection;Cisplatin Injection

INTERVENTIONS:
Drug: SHR-8068;Adebrelimab;Oxaliplatin;Capecitabine Tablets;Paclitaxel Injection;Cisplatin Injection — SHR-8068: Specified dose on specified days. Adebrelimab: Specified dose on specified days. Oxaliplatin: Specified dose on specified days. Capecitabine Tablets: Specified dose on specified days. Paclitaxel Injection: Specified dose on specified days. Cisplatin Injection: Specified dose on specified days.
  Arms: SHR-8068 combined with adebrelimab and platinum-containing chemotherapy
Drug: Adebrelimab;Oxaliplatin;Capecitabine Tablets;Paclitaxel Injection;Cisplatin Injection — Adebrelimab: Specified dose on specified days. Oxaliplatin Injection: Specified dose on specified days. Capecitabine Tablets: Specified dose on specified days. Paclitaxel Injection: Specified dose on specified days. Cisplatin Injection: Specified dose on specified days.
  Arms: Adebrelimab combined with platinum-containing chemotherapy

SUMMARY:
Objective response rate (ORR) was evaluated to evaluate the efficacy of SHR-8068 combined with adebrelimab and platinum-containing chemotherapy in first-line treatment of advanced gastric and esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to join the clinical study, and sign the informed consent, compliance is good, can cooperate with follow-up;
2. Aged 18-75 at the time of signing the informed consent;
3. Histologically or cytologically confirmed, unresectable, advanced or recurrent/metastatic adenocarcinoma of the gastric or gastroesophageal junction, or unresectable or recurrent/metastatic esophageal squamous cell carcinoma without radical chemoradiation;
4. At least one measurable lesion consistent with RECIST v1.1;
5. ECOG PS score: 0-1;
6. The organ function level is good;

Exclusion Criteria:

1. Her2-positive patients;
2. Untreated (radiation or surgery) central nervous system metastasis, or accompanied by meningeal metastasis, spinal cord compression, etc.;
3. Uncontrolled pleural effusion, pericardial effusion, or peritoneal effusion with clinical symptoms;
4. Previous or co-existing malignant neoplasms;
5. The presence of any active or known autoimmune disease;
6. People who have previously received an organ transplant;
7. Have clinical symptoms or diseases of the heart that are not well controlled;
8. Known allergic reactions to adebrelimab or other monoclonal antibodies or investigational drugs;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR based on RECIST v1.1 assessment. | All enrolled subjects were evaluated every 6 or 9 weeks starting with the first dose, up to 1 years

SECONDARY OUTCOMES:
DCR based on RECIST v1.1 assessment | All enrolled subjects were evaluated every 6 or 9 weeks starting with the first dose, up to 1 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided